CLINICAL TRIAL: NCT05355610
Title: Objective Vestibular Evaluation & Rehabilitation With Intratympanic Dexamethasone and Gentamicin in Meniere's Disease
Brief Title: Vestibular Rehabilitation With Intratympanic Drug Therapy in Meniere's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Combined Military Hospital Quetta (Other)
Responsible Party: Principal Investigator, Dr Zeeshan Ayub, Associate Professor ENT, Combined Military Hospital Quetta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: File No: CMH QTA-IRB/043
Record Dates: First submitted 2022-04-24; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Vestibular Disorder Preservation
Keywords: dexamethasone, gentamicin
MeSH Terms: interventions — Gentamicins; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients with unilateral Meniere's disease with intractable vertigo will be administered two doses of intratympanic gentamicin plus dexamethasone 1 week apart
Masking Description: For Alleviation of Intractable symptoms of Meniere's disease will be treated with intratympanic steroids. Measured with pre and post therapy vestibular severity index.
  At the same time intratympanic dexamethasone will be used to rescue hearing measured with speech reception threshold and speech discrimination threshold
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibular severity index improvement (Experimental): Improvement in vestibular symptoms with intratympanic gentamicin
  Interventions: Drug: Gentamicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Gentamicin — Intratympanic gentamicin and dexamethasone administered in two doses one week apart
  Other Names: Intratympanic gentamicin
Drug: Dexamethasone — Intratympanic gentamicin and dexamethasone administered in two doses one week apart
  Other Names: Intratympanic dexamethasone

SUMMARY:
Intractable symptoms of Meniere's disease will be treated with intratympanic steroids.

At the same time intratympanic dexamethasone will be used to rescue hearing

DETAILED DESCRIPTION:
For Alleviation of Intractable symptoms of Meniere's disease will be treated with intratympanic steroids. Measured with pre and post therapy vestibular severity index.

At the same time intratympanic dexamethasone will be used to rescue hearing measured with speech reception threshold and speech discrimination threshold

ELIGIBILITY:
Inclusion Criteria:

* All patients of unilateral Meniere's disease with severe vestibular symptoms

Exclusion Criteria:

* Bilateral disease, operated cases

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Vestibular Rehabilitation | Three months
  Improvement in vestibular severity index

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Ayub, FCPS, Principal Investigator — CMH Quetta; Zeeshan Ayub, FCPS, Study Chair — CMH Quetta
Locations (1):
- CMH Quetta, Quetta, Balochistan, Pakistan